CLINICAL TRIAL: NCT05987241
Title: MODERN: An Integrated Phase 2/3 and Phase 3 Trial of MRD-Based Optimization of ADjuvant ThErapy in URothelial CaNcer
Brief Title: Testing the Role of DNA Released From Tumor Cells Into the Blood in Guiding the Use of Immunotherapy After Surgical Removal of the Bladder, Kidney, Ureter, and Urethra for Urothelial Cancer Treatment, MODERN Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-05980; NCI-2023-05980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A032103 (Other: Alliance for Clinical Trials in Oncology); A032103 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-08-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma; Muscle Invasive Renal Pelvis Urothelial Carcinoma; Muscle Invasive Ureter Urothelial Carcinoma; Muscle Invasive Urethral Urothelial Carcinoma; Stage II Bladder Urothelial Carcinoma AJCC v6 and v7; Stage III Bladder Urothelial Carcinoma AJCC v6 and v7; Stage IV Bladder Urothelial Carcinoma AJCC v7
MeSH Terms: interventions — Specimen Handling; Cell-Free Nucleic Acids; Circulating Tumor DNA; Cystoscopy; Magnetic Resonance Spectroscopy; Nivolumab; relatlimab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A, Arm I (nivolumab) (Active Comparator): Patients in Cohort A, Arm I receive nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystoscopy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Questionnaire Administration
- Cohort A, Arm II (nivolumab, relatlimab) (Experimental): Patients in Cohort A, Arm II receive nivolumab IV over 30 minutes and relatlimab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystoscopy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Questionnaire Administration; Biological: Relatlimab
- Cohort B, Arm III (nivolumab) (Active Comparator): Patients in Cohort B, Arm III receive nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Questionnaire Administration
- Cohort B, Arm IV (ctDNA surveillance, nivolumab) (Experimental): Patients in Cohort B, Arm IV undergo ctDNA surveillance consisting of collection of tissue and blood during screening and collection of blood only on study and during follow up. Patients who convert to ctDNA(+) during surveillance then receive nivolumab IV over 30 minutes and relatlimab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: cfDNA or ctDNA Measurement; Procedure: Computed Tomography; Procedure: Cystoscopy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue and blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: cfDNA or ctDNA Measurement — Undergo ctDNA surveillance
  Other Names: Cell-Free DNA/Circulating Tumor DNA Measurement; cfDNA/ctdDNA Measurement; cfDNA/ctDNA; cfDNA/ctDNA Measurement; Circulating Cell-Free DNA/Circulating Tumor-Derived DNA Measurement
  Arms: Cohort B, Arm IV (ctDNA surveillance, nivolumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Cystoscopy — Undergo cystoscopy
  Other Names: CS
  Arms: Cohort A, Arm I (nivolumab); Cohort A, Arm II (nivolumab, relatlimab); Cohort B, Arm IV (ctDNA surveillance, nivolumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Other: Questionnaire Administration — Ancillary studies
Biological: Relatlimab — Given IV
  Other Names: BMS 986016; BMS-986016; BMS986016; Immunoglobulin G4, Anti-(human Lymphocyte Activation Gene-3 Protein) (Human Heavy Chain), Disulfide with Human Light Chain, Dimer
  Arms: Cohort A, Arm II (nivolumab, relatlimab)

SUMMARY:
This phase II/III trial examines whether patients who have undergone surgical removal of bladder, kidney, ureter or urethra, but require an additional treatment called immunotherapy to help prevent their urinary tract (urothelial) cancer from coming back, can be identified by a blood test. Many types of tumors tend to lose cells or release different types of cellular products including their DNA which is referred to as circulating tumor DNA (ctDNA) into the bloodstream before changes can be seen on scans. Health care providers can measure the level of ctDNA in blood or other bodily fluids to determine which patients are at higher risk for disease progression or relapse. In this study, a blood test is used to measure ctDNA and see if there is still cancer somewhere in the body after surgery and if giving a treatment will help eliminate the cancer. Immunotherapy with monoclonal antibodies, such as nivolumab and relatlimab, can help the body's immune system to attack the cancer, and can interfere with the ability of tumor cells to grow and spread. This trial may help doctors determine if ctDNA measurement in blood can better identify patients that need additional treatment, if treatment with nivolumab prolongs patients' life and whether the additional immunotherapy treatment with relatlimab extends time without disease progression or prolongs life of urothelial cancer patients who have undergone surgical removal of their bladder, kidney, ureter or urethra.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the ctDNA clearance proportion (i.e., ctDNA positive [+] --> ctDNA negative [-]) at 12 weeks in patients enrolled in Cohort A treated with adjuvant nivolumab versus nivolumab + relatlimab (phase 2 portion).

II. To compare overall survival in patients enrolled in Cohort A treated with adjuvant nivolumab versus nivolumab + relatlimab (phase 3 portion).

III. To compare disease-free survival in patients enrolled in Cohort B randomized to immediate treatment with nivolumab to those randomized to surveillance with subsequent treatment with nivolumab only upon converting to ctDNA(+)

SECONDARY OBJECTIVES:

I. To compare disease-free survival in patients enrolled in Cohort A treated with adjuvant nivolumab versus nivolumab + relatlimab.

II. To define the association between ctDNA clearance and disease-free survival and overall survival for Cohort A patients.

III. To compare overall survival in patients enrolled in Cohort B randomized to immediate treatment with nivolumab to those randomized to surveillance with subsequent treatment with nivolumab only upon converting to ctDNA(+).

IV. To determine the lead time from a ctDNA(+) assay to radiographic recurrence in patients initially ctDNA(-) post-definitive surgery enrolled in Cohort B.

V. To estimate the proportion of Cohort B patients on Arm 4 who become ctDNA(+) and receive nivolumab.

VI. To compare the cumulative incidence of Cohort B patients who become ctDNA(+) between Arms 3 and 4.

VII. To determine the safety of adjuvant nivolumab plus relatlimab. VIII. To compare disease-free survival and overall survival in patients enrolled in Cohort A treated with adjuvant nivolumab versus nivolumab + relatlimab according to receipt of neoadjuvant immune checkpoint blockade-containing therapy versus no neoadjuvant immune checkpoint blockade-containing therapy.

IX. To compare disease-free survival and overall survival in patients enrolled in Cohort B treated with adjuvant nivolumab versus nivolumab + relatlimab according to receipt of neoadjuvant immune checkpoint blockade-containing therapy versus no neoadjuvant immune checkpoint blockade-containing therapy.

EXPLORATORY OBJECTIVES:

I. To explore the kinetics of quantitative ctDNA levels (mean number of tumor molecules observed per mL of plasma or MTM/ml) over time and the association between ctDNA kinetics and time-to-event outcomes.

II. To estimate the costs and value of care in patients with a ctDNA(+) assay post-radical surgery treated with adjuvant nivolumab versus nivolumab + relatlimab.

III. To estimate the costs and value of care in patients with a ctDNA(-) assay post-radical surgery treated with adjuvant nivolumab versus surveillance with subsequent treatment with nivolumab at the time of conversion to ctDNA(+).

QUALITY OF LIFE OBJECTIVES:

I. Within each cohort, to compare quality-adjusted survival among randomized arms using European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L).

II. Within Cohort B, to compare overall quality of life (QOL) as measured by the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) between baseline and 42 months (calculated as the area under the curve) among randomized arms.

III. Within each cohort, to compare overall QOL as measured by the EORTC QLQ-C30 at each time point among randomized arms.

IV. Within each cohort, to compare bladder cancer-specific QOL as measured by the EORTC Bladder Cancer Muscle-Invasive 30 Questionnaire (QLQ-BLM30) at each time point among randomized arms.

V. Within each cohort, to compare patient-reported fatigue as measured by Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue at each time point among randomized arms.

OUTLINE: Patients are assigned to 1 of 2 cohorts based on ctDNA results.

COHORT A: Patients who are ctDNA(+) are randomized to 1 of 2 arms:

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and may undergo cystoscopy throughout the trial.

ARM II: Patients receive nivolumab IV over 30 minutes and relatlimab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.

COHORT B: Patients who are ctDNA(-) are randomized to 1 of 2 arms:

ARM III: Patients receive nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.

ARM IV: Patients undergo ctDNA surveillance consisting of collection of tissue and blood during screening and collection of blood only on study and during follow up. Patients who convert to ctDNA(+) during surveillance then receive nivolumab IV over 30 minutes and relatlimab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of tissue during screening and collection of blood throughout the trial. Patients also undergo CT or MRI and may undergo cystoscopy throughout the trial.

After completion of study treatment, patients are followed up at weeks 60, 72, 84, 96, 120, 144, 196, and 248.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Histologically confirmed muscle-invasive urothelial carcinoma of the urethra, bladder, ureter or renal pelvis
* PRE-REGISTRATION: Variant histology, including neuroendocrine differentiation, sarcomatoid, micropapillary, glandular, trophoblastic, Mullerian, is allowed if urothelial cancer is predominant histology (any amount of squamous differentiation is allowed provided the tumor is not a pure squamous cell cancer)
* PRE-REGISTRATION: Patient must have had radical surgery (i.e., cystectomy and lymph node dissection or nephroureterectomy or ureterectomy) ≥ 3 weeks, but ≤ 12 weeks prior to pre-registration. Patients who have had a partial cystectomy as definitive therapy are not eligible
* PRE-REGISTRATION: No gross cancer at the surgical margins. Microscopic invasive urothelial carcinoma at the surgical margins (i.e., "positive margins") are allowed. Carcinoma in situ (CIS) at margins is considered negative margins
* PRE-REGISTRATION: No evidence of residual cancer or metastasis after radical cystectomy or nephroureterectomy or ureterectomy (imaging is not required prior to pre-registration but is required prior to registration)
* PRE-REGISTRATION: Have undergone a radical cystectomy nephroureterectomy, or ureterectomy with pathological evidence of urothelial carcinoma at high risk of recurrence as described in one of the two scenarios below (i or ii). The 7th edition of American Joint Committee on Cancer (AJCC) staging will be utilized.:

  * (i) Patients who have not received neoadjuvant systemic therapy: pT3-pT4* or pT0/x-pT4/N+ on radical surgery (i.e., cystectomy, nephroureterectomy, or ureterectomy) and are not eligible for adjuvant cisplatin chemotherapy

    * (i) Patients ineligible for cisplatin due to at least one of the following criteria and reason for ineligibility should be documented:

      * (i) Creatinine Clearance (using Cockcroft-Gault): < 60 mL/min
      * (i) Common Terminology Criteria for Adverse Events (CTCAE) version 5, grade >= 2 audiometric hearing loss
      * (i) CTCAE version 5, grade >= 2 or above peripheral neuropathy
      * New York Heart Association Class III heart failure
      * (i) Eastern Cooperative Oncology Group (ECOG) performance status = 2
    * (i) Patients who are eligible for cisplatin may be candidates if they refuse adjuvant cisplatin-based chemotherapy, despite being informed by the investigator about the treatment options. The patient's refusal must be documented.

      * (i) Patients with pT2N0 urothelial cancer on radical surgery specimen (without prior neoadjuvant systemic therapy) with ctDNA(+) Signatera results based on an assay performed post-radical surgery as part of routine care outside of the study may proceed with pre-registration but require confirmation of ctDNA(+) Signatera testing on repeat "central testing" in the context of A032103 testing. Patients with pT2N0 with central testing not confirming ctDNA(+) will not be eligible for A032103 (Note: this is distinct from patients with ypT2N0 who are eligible based on ii).
  * (ii) Patients who received neoadjuvant systemic therapy: ypT2-T4a and/or ypN+ on radical surgery (i.e., cystectomy. , nephroureterectomy, or ureterectomy) pathology specimen. Neoadjuvant systemic therapy may have included cisplatin-based chemotherapy, cisplatin-based chemotherapy plus PD-1/PD-L1 blockade, or enfortumab vedotin plus PD-1/PD-L1 blockade
* PRE-REGISTRATION: Available tumor tissue for central Signatera testing to be submitted at pre-registration. Central testing is defined as testing performed as part of the A032103 study prior to registration and is provided by the study and not routine standard commercial testing. Patients who have already had local Signatera testing performed as part of routine care will require repeat central testing as part of the A032103 study to be eligible for registration/randomization. Tumor tissue from the radical surgery specimen is preferred over tissue from prior diagnostic biopsy specimen (e.g., transurethral resection of bladder tumor specimen)
* PRE-REGISTRATION: Age >= 18 years
* PRE-REGISTRATION: ECOG Performance Status 0-2
* PRE-REGISTRATION: Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects
* PRE-REGISTRATION: No postoperative/adjuvant systemic therapy after radical surgery
* PRE-REGISTRATION: No adjuvant radiation after radical surgery
* PRE-REGISTRATION: No treatment with any other type of investigational agent =< 4 weeks before pre-registration
* PRE-REGISTRATION: Not have ever received prior treatment with LAG-3 blockade
* PRE-REGISTRATION: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* PRE-REGISTRATION: Absolute Neutrophil Count (ANC) >= 1,200/mm^3
* PRE-REGISTRATION: Platelet count >= 100,000/mm^3
* PRE-REGISTRATION: Hemoglobin >= 8 g/dL
* PRE-REGISTRATION: Creatinine =< 1.5 x upper limit of normal (ULN) or calculated (calc.) creatinine clearance > 30 mL/min (using either Cockcroft-Gault formula or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* PRE-REGISTRATION: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN
* PRE-REGISTRATION: Total bilirubin =< 1.5 x upper limit of normal (ULN) (except in patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* PRE-REGISTRATION: For women of childbearing potential only: A negative urine or serum pregnancy test done =< 14 days prior to pre-registration is required
* PRE-REGISTRATION: Not currently requiring hemodialysis
* PRE-REGISTRATION: No current or prior history of myocarditis
* PRE-REGISTRATION: No grade ≥ 3 immune related adverse event with prior PD-1/PD-L1 blockade
* PRE-REGISTRATION: No active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens- Johnson syndrome, or phospholipid syndrome because of the risk of recurrence or exacerbation of disease.
* PRE-REGISTRATION: Patients with vitiligo, endocrine deficiencies including type I diabetes mellitus, thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible.
* PRE-REGISTRATION: Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* PRE-REGISTRATION: No current pneumonitis or prior history of non-infectious pneumonitis that required steroids within the previous 5 years.
* PRE-REGISTRATION: No known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* PRE-REGISTRATION: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* PRE-REGISTRATION: Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible.
* PRE-REGISTRATION: No concurrent antineoplastic therapy.
* PRE-REGISTRATION: No current immunosuppressive agents (with the exception of corticosteroids as described below).
* PRE-REGISTRATION: No condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of pre-registration (with the exception of steroid pre-medications for contrast allergies). Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* REGISTRATION: Patient must have had radical cystectomy and lymph node dissection or nephroureterectomy or ureterectomy =< 18 weeks prior to registration.
* REGISTRATION: Must have evaluable ctDNA Signatera assay result (i.e., ctDNA[+]or ctDNA[-]) based on test performed as part of central testing at pre-registration to A032103. Central testing is defined as testing performed as part of the A032103. Local/commercial testing results may not be used for registration to A032103

  * Cisplatin-ineligible (or cisplatin-declining) patients with a pT2N0 urothelial cancer on cystectomy or nephroureterectomy or ureterectomy who were pre-registered based on routine standard care ctDNA(+) Signatera testing must have confirmed ctDNA(+) Signatera testing on central testing. If central Signatera testing yields a ctDNA(-) result, these patients are ineligible. NOTE: This is a distinct consideration from patients with ypT2-4 and/or ypN+ urothelial cancer (i.e., patients who had received neoadjuvant cisplatin-based chemotherapy) who are eligible with either ctDNA(+) or ctDNA(-) central Signatera testing
* REGISTRATION: All patients must have confirmed disease-free status defined as no measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, or definitive non-measurable radiographic metastatic disease, within 60 days prior to registration. Patients with equivocal nodes less than 15 mm in short axis, or < 10 mm in long axis for non-lymph node lesions, not considered by the investigator to represent malignant disease will be eligible. Attempts should be made to resolve the etiology of equivocal lesions with complementary imaging (e.g., PET scan) or biopsy.
* REGISTRATION: No major surgery =< 3 weeks before registration.
* REGISTRATION: No live vaccine within 30 days prior to registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette- Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist [registered trademark]) are live attenuated vaccines and are not allowed. Coronavirus disease 2019 (COVID-19) vaccines are not live vaccines and are allowed
* REGISTRATION: No change since registration in clinical condition and/or laboratory tests that would impact the safety of nivolumab +/- relatlimab administration in the opinion of the treating investigator
* COHORT B, ARM 4 PATIENTS INITIATING NIVOLUMAB AFTER CONVERSION OF ctDNA ASSAY FROM ctDNA(-) to ctDNA (+):

  * Patient must have converted to ctDNA(+) during serial monitoring performed centrally in the setting of the A032103 study
* COHORT B, ARM 4 PATIENTS INITIATING NIVOLUMAB AFTER CONVERSION OF ctDNA ASSAY FROM ctDNA(-) to ctDNA (+):

  * No evidence of metastatic disease on the most recent scheduled imaging assessment as outlined in the study calendar (no repeat imaging is necessary specifically at the time of the conversion from ctDNA[-] to ctDNA[+]).
* COHORT B, ARM 4 PATIENTS INITIATING NIVOLUMAB AFTER CONVERSION OF ctDNA ASSAY FROM ctDNA(-) to ctDNA (+):

  * No change in clinical condition and/or laboratory tests that would impact the safety of nivolumab administration in the opinion of the treating investigator
* COHORT B, ARM 4 PATIENTS INITIATING NIVOLUMAB AFTER CONVERSION OF ctDNA ASSAY FROM ctDNA(-) to ctDNA (+):

  * =< 6 weeks from reporting of ctDNA(+) result to site (not from the date sample was drawn).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2030-09-02 (Estimated); Study Completion 2030-09-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are circulating tumor DNA negative (ctDNA[-]) (Cohort A Phase II) | At week 12 from treatment start date
  Will be determined for each treatment arm as the number of patients who are ctDNA(-) after 12 weeks of treatment divided by the total number of patients on the treatment arm. Patients who do not have a 12-week ctDNA result will be deemed to be ctDNA(+). The comparison of the proportions of patients who are ctDNA(-) after 12 weeks of treatment between the two arms will be performed with a chi-square test.
Overall survival (OS) (Cohort A Phase III) | From randomization until death due to any cause, assessed up to 5 years after completion of study treatment
  The analysis will be performed using a stratified log-rank test that uses the specified stratification variables. An additional analysis will be perform using a stratified Cox regression model to generate the point estimate and 90% confidence interval for the hazard ratio (HR) (comparing Arm 2 to Arm 1).
Disease-Free Survival (DFS) (Cohort B) | From randomization until confirmed disease recurrence as assessed by the treating physician or death due to any cause, assessed up to 5 years after completion of study treatment
  A stratified Cox model (using the randomization stratification variables will be used to generate a 90% confidence interval (CI) for the HR. If the 90% CI does not contain 1.39, Arm 4 (surveillance with ctDNA serial testing to determine whether patient is treated with nivolumab) will be deemed to be non-inferior to treating patients immediately with nivolumab.

SECONDARY OUTCOMES:
Proportion of patients who are ctDNA(-) (Cohort A Phase III) from treatment start date | At week 12
  Will be determined for each treatment arm as the number of patients who are ctDNA(-) after 12 weeks of treatment divided by the total number of patients on the treatment arm. Patients who do not have a 12-week ctDNA result will be deemed to be ctDNA(+).
OS (Cohort A Phase II) | From randomization until death due to any cause, assessed up to 5 years after completion of study treatment
  If the trial does not continue to phase III, OS will be a secondary endpoint.
DFS (Cohort A Phase II or III) | From randomization until confirmed disease recurrence as assessed by the treating physician or death due to any cause, assessed up to 5 years after completion of study treatment
  This will be a secondary endpoint for the phase III trial, if completed, or for the phase II trial if the phase III trial is not performed.
Incidence of adverse events (Cohort A) | Up to 5 years after completion of study treatment
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Adverse events (AEs) will be summarized with frequencies and relative frequencies. The maximum grade for an AE will be recorded for each patient by treatment arm. The number (percent) of patients that experience each observed adverse event will be summarized by treatment arm. In addition, the proportion of patients that experience a grade 3+, grade 4+, and grade 5 adverse event will be summarized as the number and percent of patients by treatment arm. The primary summary will be regardless of attribution.
OS (Cohort B) | From randomization until death due to any cause, assessed up to 5 years after completion of study treatment
Cumulative incidence of ctDNA(+) conversion (Cohort B) | From randomization until a patient becomes ctDNA(+), assessed up to 5 years after completion of study treatment
Lead time for ctDNA(+) conversion (Cohort B) | From when a patient becomes ctDNA(+) until a confirmed radiographic disease recurrence, assessed up to 5 years after completion of study treatment
Incidence of adverse events (Cohort B) | Up to 5 years after completion of study treatment
  Will be assessed using CTCAE v5.0. Adverse events will be summarized with frequencies and relative frequencies. The maximum grade for an AE will be recorded for each patient by treatment arm. The number (percent) of patients that experience each observed adverse event will be summarized by treatment arm. In addition, the proportion of patients that experience a grade 3+, grade 4+, and grade 5 adverse event will be summarized as the number and percent of patients by treatment arm. The primary summary will be regardless of attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Galsky, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (485):
- United States (477):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford HealthCare - Avon, Avon, Connecticut
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Hartford Healthcare - Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Hartford HealthCare - Manchester, Manchester, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Malcom Randall Veterans Administration Medical Center, Gainesville, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Unity Park Ridge Campus, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Cancer Center Southpoint, Durham, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Levine Cancer Institute - Huntersville, Huntersville, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Levine Cancer Institute - Union West, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Waterloo Regional Health Network, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm